CLINICAL TRIAL: NCT01032486
Title: An Open-Label, Multi-Center, Single Arm Study to Evaluate the Effects of Azilect® on Sleep Disturbances in Parkinson's Disease Subjects
Brief Title: Study for Rasagiline Effect on Sleep Trial(REST)in Parkinson's Disease
Acronym: PD
Status: Completed | Type: Observational
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TNC-RAS-PD/01; REST (Other: Teva)
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Parkinson's Disease
Keywords: Rasagiline; Sleep; Sleepiness; Parkinson's Disease Sleep Scale; Epworth Sleepiness Scale
MeSH Terms: conditions — Parkinson Disease; Sleepiness | interventions — rasagiline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Azilect: Subjects with a diagnosis of idiopathic Parkinson's disease eligible to Azilect® treatment based on the investigator's clinical assessment and according to the Canadian product monograph.
  Interventions: Drug: Rasagiline mesylate

INTERVENTIONS:
Drug: Rasagiline mesylate — Azilect® tablets (0.5mg or 1.0 mg) administered orally once daily
  Other Names: Rasagiline mesylate, Azilect

SUMMARY:
The main objective of this study is to evaluate the effect of Azilect® on sleep disturbances in Parkinson's Disease patients, after 2 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic Parkinson's disease.
* eligible to Azilect® treatment as per Canadian product monograph

Exclusion Criteria:

* exclusion (e.g. drug-drug interactions, contraindications, warnings and precautions) based on the Canadian product monograph.
* investigational drug within 30 days prior to study
* use of Azilect® or selegiline within 60 days prior to study
* significant medical condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a sample of participants with Parkinson's disease who will be prescribed Azilect® treatment as per Canadian product monograph in order to observe changes in sleep behaviour.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of the study in sleep disturbances as measured with the Parkinson's Disease Sleep Scale (PDSS). | 2 months

SECONDARY OUTCOMES:
Change from baseline to end of the study in daytime sleepiness as measured with the Epworth Sleepiness Scale (ESS). | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Michel Panisset, MD, Principal Investigator — André Barbeau Movement Disorders Unit, Centre Hospitalier Université de Montréal (CHUM)